CLINICAL TRIAL: NCT04714255
Title: The Efficacy of Art Intervention on Decreasing Pain and Anxiety During Intravenous Cannulation
Brief Title: Efficacy of Art Intervention on Decreasing Pain and Anxiety During Intravenous Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Sherzad Khudeida Suleman, Principal Investigator (PhD Student), University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSK
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Catheterization; Pain; Anxiety; Art; Children
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TICK-B group as Intervention group (Experimental): Pediatric patients received TICK-B as a distraction in the TICK-B group Trace Image and Coloring for Kids-Book were conducted on the children undergoing the Cannulation procedure.
  Interventions: Other: Trace Image and Coloring for Kids-Book (TICK-B)
- Standard care provided group as control group (No Intervention): Pediatric patients received standard care (routine care) in the control group.

INTERVENTIONS:
Other: Trace Image and Coloring for Kids-Book (TICK-B) — A collection of images attractive that need to be colored, created as a book called TICK-B. This book was created with the instructions and recommendations of a pediatric psychiatrist and a professional drawing teacher at a children's school.Distraction with TICK-B began 1-3 min. before the intravenous cannula procedure and lasted until the end of the procedure.
  Arms: TICK-B group as Intervention group

SUMMARY:
Peripheral Intravenous Cannulation (PIVC), one of the most common therapeutic procedures in medical care, can be difficult even for experienced medical practitioners. The pain of intravenous cannulation is considered the major limitation in pediatric clinical care. Reducing the pain of intravenous cannulation has been the motive for many investigations. Intervention methods used to reduce the distress related to painful procedures are widely recommended. The management of pain and anxiety is more essential because it may modify children's memory for procedural pain and the subsequent acceptance of later health care painful interventions. Distraction is the most studied psychological technique to relieve venipuncture-related pain and distress, with strong evidence supporting its efficacy in children.

Art therapy commonly used to reduce pain and anxiety of children's disease but was not used in reducing distress outcomes of painful procedures.

We used a collection of the image need for coloring and tracing called Trace Image and Coloring for Kids-Book (TICK-B).

The purpose of this study is to exam the effectiveness of TICK-B in decreasing pain and anxiety during cannulation.

DETAILED DESCRIPTION:
Peripheral Intravenous Cannulation (PIVC), one of the most common therapeutic procedures in medical care, can be difficult even for experienced medical practitioners. The pain of intravenous cannulation is considered the major limitation in pediatric clinical care. Reducing the pain of intravenous cannulation has been the motive for many investigations. Intervention methods used to reduce the distress related to painful procedures are widely recommended. The management of pain and anxiety is more essential because it may modify children's memory for procedural pain and the subsequent acceptance of later health care painful interventions. Distraction is the most studied psychological technique to relieve venipuncture-related pain and distress, with strong evidence supporting its efficacy in children.

Art therapy commonly used to reduce pain and anxiety of children's disease but was not used in reducing distress outcomes of painful procedures.

We used a collection of the image need for coloring and tracing called Trace Image and Coloring for Kids-Book (TICK-B).

The purpose of this study is to exam the effectiveness of TICK-B in decreasing pain and anxiety during cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 6-12 years old,
* Pediatric who needed peripheral cannulation,

Exclusion Criteria:

* Children with chronic conditions,
* impairments physical,
* Disabilities with communicating difficulties,
* Those whose parent not participated,
* Neurodevelopmental delayed, can't verbal speak, hearing or visual impairments,
* Children with coma or drowsiness,
* have to take analgesic medication for less than 6 hrs.
* history of syncope.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | Immediately after venipuncture (1-2 minutes after procedure, to mask , observer)
  Pain: The severity of pain measured by Faces Pain Scale-Revised (FPS-R): The FPS-R ranking is a 0-10 scale with the six cartoons.

SECONDARY OUTCOMES:
Fear Measure | Time Frame: Immediately after venipuncture (1-2 min.)
  The Childrens Fear Scale (CFS) is used to assess children's fear or anxiety levels. The one-item scale consists of five sex-neutral faces arranged from left to right with no fear in the center, through fear out to extreme fear.

OTHER OUTCOMES:
Pain and anxiety of children measured by parents and observe. | Time Frame: Immediately after venipuncture (1-2 minutes after procedure to mask observer
  outcomes Measured by Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Akram Atrushi, Professor, Study Chair — Duhok University; Margareta Halek, Professor, Study Director — Witten\Herdecke University
Locations (1):
- Sherzad Suleman, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No